CLINICAL TRIAL: NCT05278962
Title: Heart Failure Patients With Left Ventricular Assist Devices Being Treated With Sodium-Glucose Co-Transporter 2 Inhibitors
Brief Title: HF Patients With LVADs Being Treated With SGLT2i
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1986
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: left ventricular assist device; SGLT2i

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SGLT2i (Active Comparator): Participants will be asked to take an SGLT2i for 6 months. The SGLT2i and heart failure care will be managed according to routine care, and data will be collected from the participant's medical record.
  Interventions: Drug: SGLT2i
- No SGLT2i (Active Comparator): Participants will not be asked to take an SGLT2i. Heart failure care will be managed according to routine care, and data will be collected from the participant's medical record.
  Interventions: Other: No SGLT2i

INTERVENTIONS:
Drug: SGLT2i — empagliflozin (10 mg daily) or dapagliflozin (10 mg daily), depending on formulary coverage
  Arms: SGLT2i
Other: No SGLT2i — No SGLT2i
  Arms: No SGLT2i

SUMMARY:
The main purpose of this study is to observe outcomes of sodium-glucose co-transporter 2 inhibitors (SGLT2i) in heart failure (HF) patients with left ventricular assist devices (LVAD).

DETAILED DESCRIPTION:
The exact mechanism of cardiovascular benefit from SGLT2i continues to be the source of further research. The investigators hypothesize that heart failure patients with LVADs will similarly benefit from the SGLT2i-associated natriuresis and diuresis, which in turn reduces preload. This is further associated with reduced heart failure readmissions and right ventricular failure. Additionally, the animal models indicating reduced cardiac work and remodeling in this population may benefit these patients as one of the goals of LVAD implantation is to reduce cardiac energy expenditure and promote remodeling and recovery in these patients.

This is a prospective, randomized controlled study to assess cardiac benefit of SGLT2i in 40 consecutive patients with heart failure undergoing LVAD implantation. After routine LVAD implantation, patients will be randomized 1:1 to one of two routine care arms: management with an SGLT2i [empagliflozin 10 milligram (mg) daily or dapagliflozin 10 mg daily, based on formulary coverage] or no SGLT2i. The patient's treating physician will be able to override randomization assignment if they determine that the assignment is not in the patient's best interest. SGLT2i management (if applicable) and follow-up care will be dictated by routine care. Data will be collected from the subject's medical record for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. LVAD implantation
2. Have not already been prescribed management with an SGLT2i
3. Estimated glomerular filtration rate (eGFR) ≥ 30 milliliters(ml)/minute(min)/1.73 meter(m)2
4. Age ≥ 18 years-old
5. Able to provide informed consent

Exclusion Criteria:

1. Diagnosis of Type 1 diabetes mellitus
2. eGFR < 30 ml/min/1.73 m2
3. Age < 18 years-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in number of ramp stages needed to achieve hemodynamic optimization | 6 months
  Measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Mark Belkin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No